CLINICAL TRIAL: NCT05849662
Title: Risk Stratified Treatment for Patients With Newly Diagnosed Juvenile Myelomonocytic Leukemia: A Phase I/II Non-randomized Study of Trametinib and Azacitidine With or Without Chemotherapy (IND #164058)
Brief Title: A Phase I/II Study of Trametinib and Azacitidine for Patients With Newly Diagnosed Juvenile Myelomonocytic Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Therapeutic Advances in Childhood Leukemia Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T2020-004
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-08

CONDITIONS: Leukemia, Juvenile Myelomonocytic; JMML; JCML; Neurofibromatosis 1; CBL Syndrome
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile; Neurofibromatosis 1 | interventions — trametinib; Azacitidine; fludarabine; fludarabine phosphate; Injections; Cytarabine

STUDY DESIGN:
Intervention Model Description: Patients will be concurrently enrolled into both the lower-risk and high-risk arm starting at Dose Level 1. The rolling 6 design will be used during Phase 1 of the study to confirm the recommended Phase 2 dose, separately for the lower-risk and high-risk arm, with one possible de-escalation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lower-risk patients (Experimental): Lower-risk patients are defined as having a mutational burden of one clonal alteration AND a low DNA methylation classification.
  Interventions: Drug: Trametinib; Drug: Azacitidine
- High-risk patients (Experimental): High-risk patients are defined as having as having a mutational burden of more than one clonal alteration AND/OR an intermediate or high DNA methylation classification.
  Interventions: Drug: Trametinib; Drug: Azacitidine; Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: Trametinib — PO or NG QD Days 1-28
  For patients age < 6 years: 0.032 mg/kg/day at max dose = 2mg/day
  For patients age ≥ 6 years: 0.025 mg/kg/day at max dose = 2 mg/day
  Other Names: GSK1120212B; TMT212-NXA
Drug: Azacitidine — IV over 30 minutes Days 1-5
  Age < 1 year or weight <10kg:
  2.5 mg/kg/day
  Age ≥ 1 year and weight ≥ 10kg:
  75 mg/m2/day
  Other Names: 5-azacytidine; Vidaza
Drug: Fludarabine — IV over 30 minutes Days 6-10
  30 mg/m2/day (1mg/kg if <12 kg)
  Other Names: FLUDARA FOR INJECTION
  Arms: High-risk patients
Drug: Cytarabine — IV over 3 hours Days 6-10
  2000 mg/m2/day (67mg/kg if <12 kg)
  Other Names: Cytosine arabinoside; Ara-C; Cytosar
  Arms: High-risk patients

SUMMARY:
This clinical trial will test the safety and efficacy of combining trametinib and azacitidine in patients with juvenile myelomonocytic leukemia (JMML). Newly diagnosed lower-risk JMML patients will receive trametinib and azacitidine. High-risk JMML patients will receive trametinib, azacitidine, fludarabine, and cytarabine.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine the safety of combining trametinib with azacitidine for patients with newly diagnosed lower-risk JMML.
2. To determine the safety of combining trametinib with azacitidine (Aza), fludarabine (FLA) and cytarabine for patients with newly diagnosed high-risk JMML.

Dosing:

Patients with newly diagnosed lower-risk JMML will be treated with daily azacitidine for 5 days in combination with daily trametinib for 28 days per course for up to 12 courses. Patients with newly diagnosed high-risk JMML will be treated with daily azacitidine, fludarabine, and cytarabine for 5 days in combination with daily trametinib for 28 days per course for up to 2 courses.

ELIGIBILITY:
Inclusion Criteria:

Age

• Patients must be ≥ 1 month and ≤21 years of age at enrollment.

Diagnosis • Patients must meet the 2022 International Consensus Classification criteria for JMML. The diagnosis is made based on the following criteria:.

Clinical and hematologic features (the first 2 features are present in most cases; the last 2 are required):

* Peripheral blood monocyte count ≥ 1 × 109/L*
* Splenomegaly†
* Blast percentage in PB and BM < 20%
* Absence of BCR::ABL1

  * This monocyte threshold is not reached in approximately 7% of cases. †Splenomegaly is absent in 3% of cases at presentation.

II. Genetic studies (1 finding required):

* Somatic mutation in PTPN11‡ or KRAS‡ or NRAS‡ or RRAS or RRAS2‡
* Clinical diagnosis of neurofibromatosis type 1 or germline NF1 mutation and loss of heterozygosity of NF1 or somatic biallelic loss of NF1
* Germline CBL mutation and loss of heterozygosity of CBL, or somatic mutation(s) in CBL§

  * Germline mutations (indicating Noonan syndrome) need to be excluded. §Occasional cases with heterozygous splice site mutations.

Performance Level

* Karnofsky > 50% for patients ≥ 16 years of age
* Lansky > 50% for patients < 16 years of age.

Prior Therapy

* No prior leukemia directed therapy is permitted with the exception of:

  1. Cytoreduction with hydroxyurea can be initiated and continued for up to 24 hours prior to the start of trametinib.
  2. Cytoreduction with 6-mercaptopurine (6-MP) 6-MP can be initiated and continued for up to 72 hours prior to the start of trametinib.
  3. Intrathecal (IT) cytarabine, IT methotrexate or triple IT therapy (cytarabine, methotrexate and hydrocortisone) within 7 days of enrollment as part of a diagnostic evaluation.

     No prior hematopoietic stem cell transplant is permitted.

     Adequate Renal Function Defined as:
* Patient must have a calculated creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2 OR a normal serum creatinine based on age/gender in the chart below:

Maximum Serum Creatinine (mg/dL):

* 1 month to < 6 months old - Male: 0.4, Female 0.4
* 6 months to <1 year old - Male 0.5, Female 0.5
* 1 to < 2 years old - Male: 0.6, Female: 0.6
* 2 to < 6 years old - Male:0.8, Female: 0.8
* 6 to < 10 years old - Male: 1, Female: 1
* 10 to < 13 years old - Male: 1.2, Female: 1.2
* 13 to < 16 years old - Male: 1.5, Female: 1.4
* ≥ 16 years old - Male: 1.7, Female: 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR (Schwartz et al. J. Peds, 106:522, 1985) utilizing child length and stature data published by the CDC.

Adequate Liver Function Defined as:

* Direct bilirubin < 1.5 x upper limit of normal (ULN) for age or normal, AND alanine transaminase (ALT) < 5 x ULN for age.
* The hepatic requirements are waived for patients with known or suspected liver involvement by leukemia and will not be evaluable for hepatotoxicity. This must be reviewed and approved by the study chair or vice chair.

Adequate Cardiac Function Defined as:

* Ejection fraction of > or = to 50% by echocardiogram, OR
* Ejection fraction of > or = to 50% by radionuclide angiogram (MUGA).

Reproductive Function

* Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed within 2 weeks prior to enrollment.
* Female patients with infants must agree not to breastfeed their infants while on this study.
* Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study and for a minimum of 6 months after study treatment.

Exclusion Criteria:

* Patients cannot have a known allergy to any of the drugs used in the study.
* Patients cannot have a systemic fungal, bacterial, viral, or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment. The patient needs to be off pressors and have negative blood cultures for 48 hours.
* Patients cannot have a plan to administer non-protocol chemotherapy, radiation therapy, or immunotherapy during the study period.
* Patients cannot have significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with the protocol treatment or procedures, interfere with consent, study participation, follow up, or interpretation of study results.
* Patients cannot have a clinical or molecular diagnosis of Noonan syndrome. Note: patients with either neurofibromatosis type 1 or Casitas B-lineage lymphoma (CBL) syndrome (also known as Noonan-like syndrome), are eligible to enroll. Patients with Down syndrome are excluded from the study.
* Patient cannot have had prior use of hematopoietic growth factors, biologics (anti-neoplastic agent), or XRT.
* Patients cannot be taking any medications for treatment of left ventricular systolic dysfunction.
* Patients cannot have a history of or current evidence of retinal vein occlusion (RVO) or central serous retinopathy (CSR).
* Patients cannot have had prior use of any MEK inhibitor.

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-10-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of combining trametinib with azacitidine for patients with newly diagnosed lower-risk JMML. | At the end of the evaluation period of Cycle 1 (defined as 28 day cycle of therapy plus 30 days following the last dose of study therapy)
  The incidence of dose limiting toxicities (DLTs) after the 1st course of therapy will be measured at different dose levels.
To determine the safety of combining trametinib with azacitidine (Aza), fludarabine (FLA) and cytarabine for patients with newly diagnosed high-risk JMML. | At the end of the evaluation period of Cycle 1 (defined as 28 day cycle of therapy plus 30 days following the last dose of study therapy)
  The incidence of dose limiting toxicities (DLTs) after the 1st course of therapy will be measured at different dose levels.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio